CLINICAL TRIAL: NCT06490471
Title: A Clinical Study Evaluating the Safety and Performance of the Femom System Compared to the Standard of Care CTG for Antepartum Fetal Monitoring.
Brief Title: Femom System Compared to the Standard of Care CTG
Status: Not yet recruiting | Type: Observational
Sponsor: Biorithm Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 202404OSU01
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the safety and performance of the femom system compared to the standard of care CTG for antepartum fetal monitoring in pregnant women with singleton gestation > 32+0 weeks of pregnancy. The main questions it aims to answer are to assess the agreement between femom data collection (FHR, MHR, UA), and values measured via the standard of care used for prenatal monitoring (i.e. CTG). The secondary objective is to test concordance in clinical interpretability of femom traces and the standard of care CTG traces.

Participants will have the femom device and CTG attached to their abdomen. The femom device will be attached for about 30 minutes while they are wearing the device for the NST.

ELIGIBILITY:
Inclusion Criteria:

1. Female age between 18-50-year-old
2. Singleton pregnancy.
3. Should be at and above 32+0 weeks of pregnancy.
4. Able to speak and read English to understand and sign the Informed Consent.

Exclusion Criteria:

1. Participants with an intellectual or mental impairment.
2. Participants with a known allergy or hypersensitivity to ECG gel electrodes.
3. Known fetal cardiac or genetic abnormality.
4. Clinically unstable participants who require immediate medical care.
5. Participants with existing dependent or unequal relationships with any member of the research team, the researchers(s) and/or the person undertaking the recruitment/consent process.
6. Participants with implantable electronic devices such as pacemaker or ICD.
7. Participants with medical skin condition in the abdominal area (such as wounds, cuts in the skin, skin rash, etc.)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women with singleton gestation > 32+0 weeks of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
FHR | From 32 weeks gestation to labour
  The 95% confidence limits for the 95% limits of agreement (LoA) for FHR are within
  -10 and 10 bpm
MHR | From 32 weeks gestation to labour
  The 95% confidence limits for the 95% limits of agreement (LoA) for MHR are within
  -8 and 8 bpm
PPA | From 32 weeks gestation to labour
  The positive percentage agreement (PPA) for UA using femom with respect to Tocodynamometry (TOCO).

SECONDARY OUTCOMES:
Femom NST vs NST | From 32 weeks gestation to labour
  To test concordance in clinical interpretability of femom NST traces and the standard of care CTG traces.

IPD SHARING:
Plan to Share IPD: No